CLINICAL TRIAL: NCT05238870
Title: Prevention of Skin Damage in the Patient in Prone Position: Development of the "ProneTection" Education and Training Package and Study of Implementation Conditions in an Intensive Care Setting in Belgium and Sweden.
Brief Title: Prevention of Skin Damage in the Patient in Prone Position: Development of Education Interventions Based on a Training Needs Assessment Study.
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Collaborators: Örebro University, Sweden (Other)
Responsible Party: Sponsor
Other Study IDs: ProneTection#1
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-02

CONDITIONS: Pressure Ulcer; Skin Lesion; Acute Respiratory Distress Syndrome
Keywords: prone position; pressure ulcer; moisture-associated skin damage; medical device-related skin injury; skin tear; prone ventilation
MeSH Terms: conditions — Pressure Ulcer; Respiratory Distress Syndrome | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Clinicians (interviewees) from Ghent University Hospital, Belgium: Semi-structured interviews with clinicians
  Interventions: Other: Interviews for the needs analysis. No intervention.
- Clinicians (interviewees) from Brussels University Hospital, Belgium: Semi-structured interviews with clinicians
  Interventions: Other: Interviews for the needs analysis. No intervention.
- Clinicians (interviewees) from Orebro University Hospital, Sweden: Semi-structured interviews with clinicians
  Interventions: Other: Interviews for the needs analysis. No intervention.

INTERVENTIONS:
Other: Interviews for the needs analysis. No intervention. — To develop the education and training package, a needs-analysis is necessary. The clinicians' training needs will be established through interviews.

SUMMARY:
This is study 1 of 3 - of the overall project: The ProneTection Quality Improvement Project.

The three aims of this study, study 1 are:

1. to establish the training needs critical care clinicians have regarding prone positioning,
2. to investigate the conditions for effective implementation as in an intensive care setting,
3. to develop an education and training package (The ProneTection package) for an interdisciplinary team of clinicians on skin damage prevention of patients in the prone position

DETAILED DESCRIPTION:
Conduct a needs assessment by using semi-structured interviews with an interdisciplinary team of clinicians (Ghent University Hospital (UZ Gent), Brussels University Hospital (UZ Brussel) and several institutions in Sweden, mainly Örebro University Hospital).

Concurrently, investigate the conditions for effective implementation in a critical care facility using the same interviews and participants (interviewees).

Develop the education and training package (the ProneTection package). The ProneTection package will be based on

1. the results of our recently published gap-analysis study,
2. the needs assessment results from the interviews, keeping the optimal conditions (facilitators) in mind for successful implementation, and
3. the critical review and evaluation by eleven key opinion leaders from the established international expert panel

ELIGIBILITY:
Inclusion Criteria:

* • Clinicians (nurses, allied health professionals and doctors) working in intensive care units (ICU) are eligible to participate. This can include critical care nurses, respiratory therapists, physiotherapists etc.

and/or

* Nurses studying towards their speciality as critical care nurses. and/or
* Wound care specialists or those responsible for advising on skin damage prevention or managing skin damage/ wounds of the patient in the prone position.

and/or

• Educators / clinical training facilitators within the hospital or teaching at the university.

and/or

* Quality assurance managers or hospital managers. and
* Signed informed consent and voluntary participation.

Exclusion Criteria:

* Other than the inclusion criteria

Max Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Clinicians from the multidisciplinary team working with or responsible for the critically ill ventilated patient in the prone position.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2022-07-08 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Opinion and information regarding the training needs critical care clinicians have regarding prone positioned patients, with a specific focus on skin damage prevention. | Interviews will be conducted within 1-2 months.
  1. Information regarding the training needs critical care clinicians have regarding prone positioning,
  2. Opinions regarding the optimal conditions for effective implementation of the educational interventions in an intensive care setting,

SECONDARY OUTCOMES:
The development of an education and training package (The ProneTection package) for an interdisciplinary team of clinicians on skin damage prevention of patients in the prone position | 2-4 months
  Development of online educational materials based on evidence, training needs assessments and expert opinions.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri Beeckman, Prof, dr, Principal Investigator — University Ghent
Locations (2):
- Belgium (2):
  - UZ Gent, Ghent, Oost-Vlaanderen
  - Universitair Ziekenhuis Brussel, Jette

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fourie A, Ahtiala M, Black J, Hevia H, Coyer F, Gefen A, LeBlanc K, Smet S, Vollman K, Walsh Y, Beeckman D. Skin damage prevention in the prone ventilated critically ill patient: A comprehensive review and gap analysis (PRONEtect study). J Tissue Viability. 2021 Nov;30(4):466-477. doi: 10.1016/j.jtv.2021.09.005. Epub 2021 Sep 23. PMID 34583874